CLINICAL TRIAL: NCT01955590
Title: A Randomized Controlled Trial of Metacognitive Therapy and Eye Movement Desensitization and Reprocessing for Posttraumatic Stress Disorder
Brief Title: A Randomized Controlled Trial of Metacognitive Therapy and EMDR for Posttraumatic Stress Disorder
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Norwegian University of Science and Technology (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: PTSD-NTNU-1
Record Dates: First submitted 2013-09-24; First posted 2013-10-07 (Estimated); Last update posted 2019-04-03 (Actual); Status verified 2018-04

CONDITIONS: Posttraumatic Stress Disorder
Keywords: Metacognitive therapy; Eye Movement Desensitization Reprocessing (EMDR); Cognitive therapy
MeSH Terms: conditions — Stress Disorders, Post-Traumatic | interventions — Eye Movement Desensitization Reprocessing; Therapeutics

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (3):
- Metacognitive therapy (Experimental): The focus of metacognitive therapy (MCT) is on metacognitive beliefs thought to underlie the development and maintenance of posttraumatic symptomatology.
  Interventions: Behavioral: Metacognitive therapy
- EMDR (Active Comparator): Eye movement desensitization reprocessing (EMDR): participant is asked to focus on trauma-related imagery, negative cognitions and body sensations while simultaneously focusing attention to a bilateral physical stimulation.
  Interventions: Behavioral: EMDR
- Treatment as usual (Active Comparator): A group of 30 patients matched for age, gender and personality disorders receiving treatment as usual (TaU) in an outpatient setting will be included as a non-randomized comparative control condition.
  Interventions: Behavioral: Treatment as usual

INTERVENTIONS:
Behavioral: Metacognitive therapy — 8-12 sessions of manualized metacognitive therapy
  Arms: Metacognitive therapy
Behavioral: EMDR — 8-12 sessions of manualized EMDR
  Arms: EMDR
Behavioral: Treatment as usual — 8-12 sessions of treatment of usual
  Arms: Treatment as usual

SUMMARY:
Posttraumatic stress disorder (PTSD) is a frequently occurring and often debilitating anxiety disorder resulting from exposure to trauma. Trauma-focused cognitive-behavioural therapies, such as Eye movement desensitization and reprocessing (EMDR), are generally considered to be evidence-based treatments for PTSD. Although a majority of patients achieve improvement, a substantial minority either drop out of treatment, present with residual symptoms following treatment or fail to make any improvement. Furthermore, a substantial portion of the clinical trials on PTSD is characterised by major methodological limitations. In addition, there's a pressing need for research on mediators of treatment outcome. Taken together, these results highlight the need for methodological rigorous and stringent clinical trials comparing treatment modalities for PTSD. The first aim of this study is to investigate whether a treatment not based on the principles of exposure, i.e. metacognitive therapy (MCT) is as efficient as exposure-based treatments. The second aim to elucidate potential mediators of treatments effects by incorporating process-related variables.

DETAILED DESCRIPTION:
EMDR is based on the assumption that posttraumatic symptoms are due to the traumatic experience(s) being stored in an unprocessed way disconnected from existing memory networks. The procedure in EMDR is postulated to facilitate the processing of the traumatic memory into existing memory networks. There is currently no empirical knowledge as to the therapeutic mechanisms of EMDR, but the protocol overlaps with core components of cognitive behavior therapy (CBT), such as imaginal exposure and cognitive restructuring of negative trauma-related cognitions. Thus, EMDR could be viewed as a form of CBT, although its originator maintains that it is a distinct treatment. EMDR is usually considered an evidence-based treatment of PTSD.

MCT is one of the new approaches in the treatment of PTSD. The metacognitive model posits that adaptation following exposure to trauma depends on metacognitive beliefs that guide how the individual interprets and responds to posttraumatic symptoms and can lead to styles of thinking that facilitate or impede emotional processing. MCT focuses on "unlocking" or removing the barriers to natural adaptation. This equips the client with general skills and therefore protects the individual from the risk of any future re-traumatisation. In contrast to EMDR, MCT does not involve proscribed exposure exercises or restructuring of negative trauma-related cognitions.

In addition we will include a group of 30 patients matched for age, gender and personality disorders receiving treatment as usual (TaU) in an outpatient setting as a non-randomized comparative control condition.

ELIGIBILITY:
Inclusion Criteria:

* a primary diagnosis of PTSD according to the Anxiety Disorders Interview Schedule (ADIS-IV)
* not previously received EMDR or MCT for this diagnosis
* not actively suicidal, presenting with suicidal ideation, psychotic or suffering from severe depression
* no evidence of alcohol or drug dependence
* Symptom chronicity of >3 months post-trauma

Exclusion Criteria:

* PTSD is not the primary diagnosis
* expressing suicidal ideation, actively psychotic, or engaging in overt self-harm
* Evidence of alcohol or drug dependence requiring treatment in its own right
* Borderline personality disorder
* Symptom chronicity <3 months post-trauma
* no ability to understand or speak Norwegian

Min Age: 16 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 96 (Actual)
Dates: Start 2012-11 (Actual); Primary Completion 2017-12 (Actual); Study Completion 2019-03-15 (Actual)

PRIMARY OUTCOMES:
Posttraumatic Stress Disorder Scale (PDS) | 8-12 weeks post-treatment
Posttraumatic Stress Disorder Scale (PDS) | 12 month follow-up

SECONDARY OUTCOMES:
Anxiety Disorders Interview Schedule (ADIS-IV) | Pre-treatment/baseline; 8-12 weeks post-treatment
PTSD Symptom Scale - Interview (PSS-I) | Pre-treatment/baseline; 8-12 weeks post-treatment
Impact of Event Scale - Revised (IES-R) | Pre-treatment/baseline; 8-12 weeks post-treatment; 12 month follow-up
Beck Anxiety Inventory (BAI) | Pre-treatment/baseline; 8-12 weeks post-treatment; 12 month follow-up
Beck Depression Inventory (BDI-II) | Pre-treatment/baseline; 8-12 weeks post-treatment; 12 month follow-up
Metacognitions Questionnaire - 30 (MCQ-30) | Pre-treatment/baseline; weekly; 8-12 weeks post-treatment
  Process outcome / mediator measure
Posttraumatic Cognitions Inventory (PTCI) | Pre-treatment/baseline; weekly; 8-12 weeks post-treatment
  Process outcome / mediator measure
Session Rating Scale (SRS) | Pre-treatment/baseline; weekly; 8-12 weeks post-treatment
  Process outcome / mediator measure
Inventory of Interpersonal Problems (IIP-64-C) | Pre-treatment/baseline; 8-12 weeks post-treatment; 12 month follow-up
Posttraumatic Stress Disorder Scale (PDS) | Weekly
WHO-5 Well-Being Index | Pre-treatment/baseline; 8-12 weeks post-treatment; 12 month follow-up

OTHER OUTCOMES:
Posttraumatic Stress Disorder Scale (PTSD-S) | Pre-treatment/baseline; weekly; 8-12 weeks post-treatment
  Only administered in the MCT treatment arm

CONTACTS AND LOCATIONS:
Overall Officials: Hans M Nordahl, Prof, Study Director — Department of Psychology, Norwegian University of Science and Technology
Locations (1):
- Outpatient speciality clinic for PTSD and other trauma-related emotional disorders at Østmarka, St. Olav University Hospital, Trondheim, Norway

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Nordahl HM, Halvorsen JO, Hjemdal O, Ternava MR, Wells A. Metacognitive therapy vs. eye movement desensitization and reprocessing for posttraumatic stress disorder: study protocol for a randomized superiority trial. Trials. 2018 Jan 8;19(1):16. doi: 10.1186/s13063-017-2404-7. PMID 29310718
- [Background] Nordahl HM, Halvorsen JO, Hjemdal O, Ternava MR, Wells A. Correction to: Metacognitive therapy vs. eye movement desensitization and reprocessing for posttraumatic stress disorder: study protocol for a randomized superiority trial. Trials. 2018 Mar 6;19(1):164. doi: 10.1186/s13063-018-2536-4. PMID 29510757